CLINICAL TRIAL: NCT00522938
Title: A Phase I-II, Multicenter, Open-label Trial of Co-administered CHR-2797 and Erlotinib in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer
Brief Title: Clinical Trial of the Safety and Effectiveness of CHR-2797 With Erlotinib in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Very poor recruitment of patients to the study
Sponsor: Chroma Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CHR-2797-005
Record Dates: First submitted 2007-08-29; First posted 2007-08-30 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Lung; Cancer; Non-small; Lung Cancer; NSCLC; erlotinib; oral; Locally Advanced Non-small Cell Lung Cancer; Metastatic Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Lung Neoplasms | interventions — tosedostat; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: CHR-2797 (tosedostat) — Once daily, oral ingestion of CHR-2797 capsules(PhaseI: 120mg, 160mg or 200mg depending on cohort or Phase II: recommended dose) capsules until progressive disease or withdrawal from the study
Drug: erlotinib — Once daily, oral ingestion of erlotinib tablets 150mg tablets until progressive disease or withdrawal from the study. Per protocol, the Investigator may reduce the dose of erlotinib or cease treatment with erlotinib(per label) with Sponsor approval.
  Other Names: Tarceva

SUMMARY:
This is an open-label, multicenter, multiple-dose, Phase I-II study of CHR-2797 co-administered with erlotinib in patients with histologically or pathologically confirmed Stage IIIB (with pleural effusion), Stage IV, or recurrent metastatic NSCLC. Throughout this protocol, "study medication" includes both CHR-2797 and erlotinib.

This study will involve 2 distinct study phases. Study Phase A will assess safety and determine the MTD of the combination of CHR-2797 and erlotinib. In addition, PK profiles for the combination of CHR-2797 and erlotinib will be evaluated. In Study Phase B, the dose chosen based on the maximum tolerated dose established in Study Phase A will be administered in a single-arm treatment design in order to evaluate the efficacy of co-administration of CHR-2797 and erlotinib.

DETAILED DESCRIPTION:
Study Phase A:

Maximum tolerated dose will be determined during Cycle 1. Tumor assessments will be made after Cycle 2 (56 days), although it is not mandatory for Phase A patients to have measurable disease. Patients who have satisfactory outcomes after Cycle 2 may continue treatment for up to a year with erlotinib 150 mg/day, and the dose of CHR-2797 they received in Study Phase A.

Study Phase B:

Patients will be treated with the dose of CHR-2797 selected in Study Phase A and 150mg/day erlotinib. Patients will receive 2 cycles of treatment (56 days) before efficacy assessment. Patients who have complete response, partial response, or stable disease are eligible to continue the study for up to a year until disease progression or unacceptable toxicity. If a patient has complete response, partial response, or stable disease at the end of the 1-year study period and the Investigator believes that continuation treatment would be beneficial, the patient may continue to be treated at the dose of CHR-2797 under a separate protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically and/or pathologically confirmed NSCLC (cytologic specimens obtained by brushing, washing, or needle aspiration of a defined lesion are acceptable). This includes the histologic subtypes of squamous cell, adeno, large cell, anaplastic cell, bronchioalveolar carcinoma, and NSCLC not otherwise specified (NOS). Note that tumors with the presence of small cell anaplastic elements are not eligible
2. NSCLC with documentation of Stage IIIB (with pleural effusion), or Stage IV, or recurrent metastatic disease based on current TNM classification
3. Disease progression or relapse following failure of platinum-based chemotherapy
4. For Study Phase A, patients are not required to have measurable disease (according to RECIST criteria) for enrollment. For patients in Study Phase B, patients must have measurable disease according to RECIST, defined by at least 1 lesion that can be accurately measured. All other lesions (e.g., pleural effusions) including small lesions (<1 cm×1 cm by spiral CT scan) are considered non-measurable for the purposes of this study. Baseline tumor measurements are to be completed as close as possible to, but no longer than 14 days before the start of study treatment
5. Prior radiation to the measurable site(s) of disease is not allowed, unless disease progression has been documented at that site since the radiotherapy. Patients who have had extensive radiotherapy are also excluded, because of the associated myelosuppressive effect
6. Prior surgery is allowed, provided it was completed at least 4 weeks prior to enrollment and the patient has recovered from surgery.
7. No known prior primary brain, metastatic brain, or meningeal tumors or clinical signs or symptoms of brain metastases
8. Able to understand and willing to sign an informed consent document
9. Age ≥18 years
10. Predicted life expectancy >3 months
11. Eastern Cooperative Oncology Group (ECOG) performance status score ≤2
12. Laboratory values within the normal or reasonable ranges and, specifically,adequate bone marrow, hepatic, and renal function including the following:

    * Hemoglobin >10 g/dL, absolute neutrophil count (ANC)>1.5×109/L, platelets ≥100×109/L
    * Total bilirubin ≤1.5× upper limit normal (ULN)
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <2.5×ULN or <5×ULN in patients with documented liver metastases
    * Creatinine ≤1.5×ULN or calculated creatinine clearance ≥60 mL/min
13. Female patients with reproductive potential must have a negative serum pregnancy test within 72 hours prior to start of study medication. All female patients of childbearing potential, and all male patients, must agree to use a medically acceptable method of contraception or agree to be abstinent throughout the treatment period and for 3 months after discontinuation of treatment. (See Section 4.1for more information.)
14. Screening for LVEF >= 55%

Exclusion Criteria:

1. Excluded therapies:

   * Concurrent anti-cancer therapy
   * Treatment with cytotoxic agents within the last 3 or 4 weeks, depending on the usual frequency of administration of the regimen, or within the last 6 weeks for agents such as mitomycin. Patients must have had resolution of acute treatment-related toxicities to baseline or National Cancer Institute Common Toxicity Criteria (NCI-CTC) Grade <1, with the exception of alopecia
   * Therapy within the last 28 days or while on study with another investigational drug
   * Use of biological response modifiers, such as granulocyte-colony stimulating factor (G-CSF) or erythropoietin, within 28 days of enrollment
   * Prior therapy with an epidermal growth factor receptor (EGFR) inhibitor
   * Radiation to the site(s) of measurable disease, unless disease progression has been documented at that site since the radiotherapy.
   * Need for palliative radiotherapy of indicator lesions
   * Treatment with known strong CYP3A4 inhibitors, for example '- azole antifungals, protease inhibitors, erythromycin, clarithromycin within 2 weeks of enrollment or at any time during the study
   * Treatment with strong CYP3A4 inducers such as rifampicin, rifabutin or rifapentine within 2 weeks of enrollment or at any time during the study
   * Warfarin or doses of coumadin (or equivalent) that are higher than 1mg/day
2. Excluded medical conditions:

   * Current hematological malignancy
   * Gastro-intestinal abnormalities including:

     * Inability to take oral medication
     * Requirement for intravenous (IV) alimentation
     * Malabsorption syndrome
     * Active peptic ulcer disease
   * A serious uncontrolled medical disorder or active infection which would impair their ability to receive study treatment
   * Known primary brain, metastatic brain, or meningeal tumors, or clinical signs or symptoms of brain metastases
   * Second malignancy (except adequately treated basal cell carcinoma of the skin or in-situ carcinoma of the cervix or breast)
   * Known history of human immunodeficiency virus (HIV) infection or chronic hepatitis B or C
   * Uncontrolled hypercalcemia (>NCI-CTC Grade 1)
   * Significant cardiovascular disease including but not limited to the following:

     * History (past or present) of congestive heart failure
     * History (past or present) of angina pectoris requiring medication
     * History of myocardial infarction with past 12 months
     * Presence of clinically significant valvular heart disease
     * History (past or present) of arrhythmia requiring treatment
     * Presence of conduction defect on Screening ECG
     * History (past or present) of uncontrolled hypertension
   * Patients with interstitial lung disease
3. Major surgery within 4 weeks prior to enrollment
4. >20% weight loss in previous 3 months
5. Pregnant or lactating women
6. Known rapidly deteriorating liver function tests (2×ULN rise in 1 week)
7. Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and/or compliance with the requirements of the protocol
8. Known or suspected allergy to any study medication used in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-12; Primary Completion 2008-02 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Study Phase A- To determine the safety, tolerability, and maximum tolerated dose (MTD) of CHR-2797 when co-administered with erlotinib | end of study
Study Phase B- To determine the objective tumor response rate to CHR-2797 and erlotinib when co-administered to patients with histologically and/or pathologically confirmed Stage IIIB, Stage IV, or recurrent metastatic non-small cell lung cancer (NSCLC) | End of study

SECONDARY OUTCOMES:
Study Phase A- To determine the pharmacokinetic (PK) profiles of CHR-2797 and erlotinib when co-administered | End of study
Study Phase B- To further evaluate the efficacy of the combination of CHR-2797 and erlotinib in patients with locally advanced or metastatic non small cell lung cancer (NSCLC) | End of study
Study Phase B- To determine the safety and tolerability of CHR-2797 and erlotinib when co administered. To determine the trough levels of CHR-2797 and erlotinib after co-administration for 28 days | End of study

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Medical Oncology Care Associates, Orange, California
  - Oncology Associates of West Kentucky, Paducah, Kentucky
  - Richmond University Medical Center, Staten Island, New York
  - Montefiore Medical Center, The Bronx, New York
  - Clinworks Research Center, Charlotte, North Carolina
  - Carolina BioOncology Institute, Huntersville, North Carolina